CLINICAL TRIAL: NCT00488579
Title: Routine Iron Prophylaxis During Pregnancy - Effects on Maternal and Child Health in Maputo City and Province (Mozambique)
Brief Title: Routine Iron Prophylaxis During Pregnancy
Acronym: PROFEG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Istitute For Health and Welfare, Finland (Other Government)
Collaborators: Academy of Finland (Other)
Responsible Party: Principal Investigator, Elina Hemminki, MD, Research Professor, THL, National Istitute For Health and Welfare, Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PROFEG
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Pregnancy
Keywords: iron prophylaxis; pregnancy; birth weight; prematurity; perinatal mortality
MeSH Terms: conditions — Birth Weight; Premature Birth; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- routine iron prophylaxis (Active Comparator): giving 60 mg ferrous sulphate daily (+folic acid)
  Interventions: Drug: Two policies of iron prophylaxis
- screening and therapy (Active Comparator): doing Hb measurement on each visit, Hb>9g/dl giving only folic acid, Hb<9g/dl giving 60-120 mg of ferrous sulphate daily (+folic acid)
  Interventions: Drug: Two policies of iron prophylaxis

INTERVENTIONS:
Drug: Two policies of iron prophylaxis — 60mg ferrous sulphate daily (+folic acid); Screening and therapy: Hb measurement on each visit, Hb>9g/dl only folic acid, Hb<9g/dl 60-120 of ferrous sulphate daily (+folic acid).

SUMMARY:
Comparison of two policies of iron administration during pregnancy in regard to health and program feasibility in an area with endemic malaria and high prevalence of HIV infection. The policies are: 1) routine iron prophylaxis, 2) screening and therapy with iron.

DETAILED DESCRIPTION:
Aim of the study:

Comparison of two policies of iron administration during pregnancy in regard to health of the mother and infant and program feasibility. The two groups compared are:

1. Routine iron prophylaxis
2. Screening of anaemia and therapy with iron

Hypothesis: group 2 will have better health outcomes.

Study groups:

Routine group: 60 mg per day of ferrous sulphate (combination with folic acid) daily.

Screening and therapy: Hb measurement on each visit, Hb >9g/dl Þ only folic acid, Hb <9g/dl Þ 60/120 mg of ferrous sulphate daily(+ folic acid)

Methods:

A pragmatic randomised controlled trial with non-blind design. Total intended sample size was 4000 women. Study site: Mozambique, Maputo City. Women are randomised individually and allocated into the two groups; 1) Routine iron prophylaxis, 2) Screening and therapy for anemia.

The recruitment of pregnant women was done in two health centres, one in Maputo city and one in Maputo Province. The women are followed in prenatal visits and until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at their first prenatal visit

Exclusion Criteria:

* Women under 18 years, high obstetric risk pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4326 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Preterm delivery | Until birth
  Birth <37 gestational weeks
Low birth weight | At birth
  weight <2500g

SECONDARY OUTCOMES:
perinatal mortality, complications during pregnancy and birth | pregnancy and neonatal period

CONTACTS AND LOCATIONS:
Overall Officials: Elina Hemminki, PhD, MD, Principal Investigator — THL; Baltazar Chilundo, Study Director — Eduardo Mondlane University
Locations (1):
- Universidade Eduardo Mondlande, Faculty of Medicine, Department of Community Health, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hemminki E, Nwaru BI, Salome G, Parkkali S, Abacassamo F, Augusto O, Cliff J, Regushevskaya E, Dgedge M, Sousa C, Chilundo B. Is selective prenatal iron prophylaxis better than routine prophylaxis: final results of a trial (PROFEG) in Maputo, Mozambique. BMJ Open. 2016 Jun 13;6(6):e011280. doi: 10.1136/bmjopen-2016-011280. PMID 27297013
- [Derived] Nwaru BI, Salome G, Abacassamo F, Augusto O, Cliff J, Sousa C, Regushevskaya E, Parkkali S, Hemminki E. Adherence in a pragmatic randomized controlled trial on prophylactic iron supplementation during pregnancy in Maputo, Mozambique. Public Health Nutr. 2015 Apr;18(6):1127-34. doi: 10.1017/S1368980014001359. Epub 2014 Jul 7. PMID 24999785
- [Derived] Parkkali S, Abacassamo F, Nwaru BI, Salome G, Augusto O, Regushevskaya E, Dgedge M, Sousa C, Cliff J, Chilundo B, Hemminki E. Comparison of routine prenatal iron prophylaxis and screening and treatment for anaemia: pregnancy results and preliminary birth results from a pragmatic randomised controlled trial (PROFEG) in Maputo, Mozambique. BMJ Open. 2013 Feb 8;3(2):e001948. doi: 10.1136/bmjopen-2012-001948. Print 2013. PMID 23396557
- [Derived] Nwaru BI, Parkkali S, Abacassamo F, Salome G, Chilundo B, Augusto O, Cliff J, Dgedge M, Regushevskaya E, Nikula M, Hemminki E. A pragmatic randomised controlled trial on routine iron prophylaxis during pregnancy in Maputo, Mozambique (PROFEG): rationale, design, and success. Matern Child Nutr. 2015 Apr;11(2):146-63. doi: 10.1111/mcn.12006. Epub 2012 Oct 1. PMID 23020829